CLINICAL TRIAL: NCT06101784
Title: A Double-Blind, Placebo-Controlled, Randomized, Adaptive, First-in-Human Study to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of Avenanthramide
Brief Title: Single and Multiple Ascending Oral Doses of Avenanthramide
Acronym: AvenActive
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Ceapro Inc. (Industry); The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROJ1602
Record Dates: First submitted 2023-08-07; First posted 2023-10-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Inflammation
Keywords: Healthy subjects; Single ascending dose; Multiple ascending dose; Natural product; Placebo controlled; First in human
MeSH Terms: conditions — Inflammation | interventions — avenanthramide-2C

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled, Randomized, Adaptive, First-in-Human Study, Single and Multiple Ascending Oral Doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Avenanthramide tablet single oral dose (Active Comparator): adaptive dose levels
  Interventions: Drug: Avenanthramide
- Placebo to match Avenanthramide tablet single oral dose (Placebo Comparator): adaptive dose levels
  Interventions: Drug: Placebo
- Avenanthramide tablet multiple oral dose (Active Comparator): adaptive dose levels
  Interventions: Drug: Avenanthramide
- Placebo to match Avenanthramide tablet multiple oral dose (Placebo Comparator): adaptive dose levels
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avenanthramide — In each cohort 6 subjects will be assigned to the active treatment and 2 subjects will be assigned to the placebo.
  Arms: Avenanthramide tablet multiple oral dose; Avenanthramide tablet single oral dose
Drug: Placebo — In each cohort 6 subjects will be assigned to the active treatment and 2 subjects will be assigned to the placebo.
  Arms: Placebo to match Avenanthramide tablet multiple oral dose; Placebo to match Avenanthramide tablet single oral dose

SUMMARY:
Avenanthramides (AVA) are di-phenolic compounds found only in oats and are of interest due to suggested bioactivities, including antioxidant and anti-inflammatory effects in vitro and in vivo.

Published data suggests that polyphenols can work as modifiers of signal transduction pathways to elicit their beneficial effects. These natural compounds express anti-inflammatory activity by modulation of pro-inflammatory gene expression such as cyclo-oxygenase, lipoxygenase, nitric oxide synthases and several pivotal cytokines, mainly by acting through nuclear factor-kappa B and mitogen-activated protein kinase signaling. The biomarkers of inflammation in blood, i.e., pro-inflammatory cytokines, chemokines, as well as other inflammatory markers (i.e., high sensitivity C-reactive protein) are of particular interest.

Primary Objectives:

* To assess the safety and tolerability of single ascending oral doses of avenanthramide in healthy subjects.
* To assess the safety and tolerability of multiple ascending oral doses of avenanthramide in healthy subjects and subjects with elevated waist circumference and low-grade inflammation.

Secondary Objectives:

* To determine the pharmacokinetics of avenanthramide following single ascending oral doses in healthy subjects.
* To compare the pharmacokinetics of avenanthramide following single oral dose in healthy subjects under fasting and fed conditions.
* To determine the pharmacokinetics of avenanthramide following multiple ascending oral doses in healthy subjects.
* To determine the pharmacokinetics of avenanthramide following multiple ascending oral doses in subjects with elevated waist circumference and low-grade inflammation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subjects;
* 2. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively, for subjects participating in Part A and Part B;
* 3. Age 18-60 years;
* 4. Willing to avoid rigorous physical activity 1 day prior to the first drug administration and during study participation;
* 5. Willing to avoid oat consumption for 1 week prior to the first drug administration and during study participation;
* 6. Non- or ex-smoker; an ex-smoker is defined as someone who completely stopped using nicotine products for at least 6 months prior to the first study drug administration;
* 7. Non- or ex-consumer of cannabis; an ex-consumer of cannabis is defined as someone who stopped using cannabis derived products for at least 6 months prior to the first study drug administration;
* 8. Have no clinically significant diseases captured in the medical history and no evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by the investigator;
* 9. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by the investigator;
* 10. Provision of signed and dated informed consent form (ICF);
* 11. Stated willingness to comply with all study procedures and availability for the duration of the study;
* 12. A male subject meeting one of the following criteria:

  1. Subject is able to procreate and agrees to use one of the accepted contraceptive regimens and not donate sperm from the first study drug administration to at least 90 days after the last drug administration. An acceptable method of contraception includes one of the following:

     * True abstinence from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject (not periodic abstinence)
     * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) If the subject has a partner of childbearing potential, he and/or his partner must agree to use two acceptable birth control methods.

     Or
  2. Subject is unable to procreate; defined as surgically sterile (i.e., has undergone a vasectomy at least 6 months prior to the first study drug administration)
* 13. A female subject meeting one of the following criteria:

  1. Subject of childbearing potential must agree to use an effective double method of birth control from the first study drug administration to at least 30 days after the last drug administration: barrier method (e.g., male or female condoms, spermicides, sponges, foams, jellies, and diaphragm) in combination with other methods of contraception including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices; or must have a sterile sexual partner.

     Or
  2. Subject is of childbearing potential and agrees to abide by true abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject (not periodic abstinence) Or
  3. Subject is of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a menopausal state (i.e., at least 1 year without menses prior to the first study drug administration).
* Part-C:

Inclusion Criteria modified:

In addition to the above criteria, the inclusion criterion #2 is defined as following:

2*. Body mass index (BMI) within 18.5 kg/m2 to 34.0 kg/m2, inclusively, for the subjects participating in Part C.

Also, subjects with elevated waist circumference and low-grade inflammation must meet the following criteria in order to be included in the study:

* Waist circumference ≥ 100 cm in men and ≥ 85 cm in women
* Hs-CRP equal or greater than 2.0 mg/L and less than 10.0 mg/L at Screening

Exclusion Criteria:

* 1. Allergy to any ingredient of the Investigational Products, including excipients;
* 2. Oat products consumption within 1-week prior the first drug administration;
* 3. History of significant hypersensitivity to any excipients of the formulation, as well as severe hypersensitivity reactions (like angioedema) to any drug;
* 4. Presence of significant gastrointestinal (GI) conditions that interfere with absorption;
* 5. Presence of significant cardiovascular disease, gastrointestinal disease, kidney disease, or endocrine disease: including diabetes, and untreated thyroid disease, or rheumatoid arthritis;
* 6. Diagnosis of Gilbert syndrome;
* 7. Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 95 mmHg at screening;
* 8. Major trauma or surgery within 3 months of study participation;
* 9. Presence of clinically significant ECG abnormalities at the screening, as defined by medical judgment;
* 10. Any clinically significant illness in the 28 days prior to the first study drug administration;
* 11. Any history of tuberculosis or proven contact with tuberculosis;
* 12. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration;
* 13. Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HbsAg (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests at screening;
* 14. Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to the first drug administration;
* 15. Use of any prescription drugs (with the exception of contraceptive or hormone replacement therapy) in the 28 days prior to the first study drug administration;
* 16. Regular use of anti-inflammatory drugs such as NSAIDs or aspirin in the 28 days prior to the first study drug administration;
* 17. Rigorous physical activity the day prior the first drug administration;
* 18. Nicotine smoking and/or nicotine replacement use;
* 19. Drinking alcohol >10 drinks/week, or history of drug abuse;
* 20. Strict dietary restrictions (such as ketogenic or vegan diet);
* 21. Regular use of nutraceuticals such as resveratrol, immune boosters, glucosamine, chondroitin, Coenzyme Q10 supplementation in the 28 days prior to the first study drug administration;
* 22. Regular use of plant concentrates (including garlic, gingko, St. John's wort) homeopathic remedies, probiotics, or fish oil (including cod liver oil), in the 28 days prior to the first drug administration;
* 23. Females who are lactating or are pregnant according to the pregnancy test at screening or prior to the first study drug administration;
* 24. Subjects who have already been included in a previous group/cohort for this clinical study;
* 25. Subjects who took an Investigational Product (IP) in the 28 days prior to the first study drug administration;
* 26. Subjects who donated 50 mL and up to 450 mL of blood in the 28 days prior to the first study drug administration;
* 27. Donation of 450 mL or more of blood (Canadian Blood Services, Hema Quebec, clinical studies, etc.) in the 2 months prior to the first study drug administration for males, and in the 3 months prior to the first drug administration for females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-12-09 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  Incidence of AEs on active treatment compared to placebo
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Alanine aminotransferase (IU/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Aspartate aminotransferase (IU/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Total bilirubin (umol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Direct bilirubin (umol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters :Indirect bilirubin (umol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Serum urea (mmol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Serum creatinine (umol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : eGFR (mL/min/1.73 mE2)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Blood urea nitrogen (mg/dL)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Fasting glucose (mmol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Fasting plasma insulin (pmol/L)
Change in laboratory parameters (general biochemistry) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters : Total cholesterol (mmol/L))
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: (Leucocytes (10E9/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Erythrocytes (10E12/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Platelets count (10E9/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Hemoglobin (g/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Hematocrit (L/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Mean corpuscular volume (fL)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Mean corpuscular hemoglobin (pg)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Mean corpuscular hemoglobin concentration (g/L)
Change in laboratory parameters (hematology) | from drug administration up to 24 hours after the last dose
  The change in serum laboratory parameters: Mean platelet volume (fL)
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: head and neck
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: cardiovascular
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: respiratory
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: abdomen
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: brief neurological appearance
Change in physical examination (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in review of body systems: brief general appearance
Change in vital signs (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in pulse rate (pbm)
Change in vital signs (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in blood pressure (mm Hg)
Change in vital signs (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in body temperature (degrees Celsius).
Change in ECG parameters (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in ECG parameters: PR interval
Change in ECG parameters (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in ECG parameters: QRS interval
Change in ECG parameters (Safety and Tolerability) | from drug administration up to 24 hours after the last dose
  The change in ECG parameters: QT interval

SECONDARY OUTCOMES:
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 on the food-effect cohort): Cmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 on the food-effect cohort): Tmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): AUC0-T
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): AUC0-∞,
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): AUC 0-T/∞
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): λz
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): T1/2
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): CL/F*
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD])
  Plasma Day 1 (and Day 8 for food effect only): VD/F*
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD]):
  Urine Day 1 (and Day 8 on the food-effect cohort): Ae
  *for parent drug only:
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD]):
  Urine Day 1 (and Day 8 on the food-effect cohort): Fe*
  *for parent drug only:
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part A (Single Ascending Dose [SAD]):
  Urine Day 1 (and Day 8 on the food-effect cohort): Clr*
  *for parent drug only:
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 1: Cmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 1: Tmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 1: AUC0-12
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Days 2 (prior to AM and PM dose), and 3 (prior to AM dose): Ctrough
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: Cmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: Tmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: Cmin
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: AUC0-24
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: AUCtau
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: T1/2
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: Rac(Cmax)
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Plasma Day 3: Rac(AUC)
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Urine Day 1 (12hrs), Day 3 (12hrs and 24hrs): Ae
  * for parent drug only
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Urine Day 1 (12hrs), Day 3 (12hrs and 24hrs): Fe*
  * for parent drug only
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part B (Multiple Ascending Dose [MAD]) in healthy subjects:
  Urine Day 1 (12hrs), Day 3 (12hrs and 24hrs): Clr*
  * for parent drug only
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 1: Cmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 1: Tmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 1: AUC0-12
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Days 8, 15, 22 and 29 (prior to AM dose): Ctrough
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : Cmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : Tmax
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : Cmin
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : AUC0-24
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : AUCtau
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : T1/2
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : Rac(Cmax)
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Plasma Day 29 : Rac(AUC)
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Urine Day 1 (12hrs) and Day 29 (12hrs and 24hrs). Ae
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Urine Day 1 (12hrs) and Day 29 (12hrs and 24hrs). Fe*
The change in Pharmacokinetics | Up to 24 hours after the last dose
  Part C (MAD in subjects with elevated waist circumference and low-grade inflammation):
  Urine Day 1 (12hrs) and Day 29 (12hrs and 24hrs). Clr*

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada